CLINICAL TRIAL: NCT02210299
Title: TEXTO : Total EXposure To Organic Pollutants
Acronym: TEXTO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Rennes University Hospital (Other)
Collaborators: Institut de Recherche en Santé, Environnement et le Travail, France (Other); Laboratoire d'Etude des Résidus et Contaminants dans les Aliments (Unknown); Institut national de l'environnement industriel et des risques (Industry); National Agency for Sanitary Safety of the Food of the Environment and Labor (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 35RC13_8917_TEXTO; 2014-A00782-45 (Other: ID RCB); 14/25-941 (Other: CPP); 140682B-82 (Other: ANSM)
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: Healthy young children (2-6 months ; 12-18 months)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exposure study (Other): 2-6 months-old children and 12-18 months-old children
  Interventions: Other: Exposure study

INTERVENTIONS:
Other: Exposure study — Sampling of blood, food, water, air and dust and delivery of dietary questionnaire

SUMMARY:
People are, especially in industrialized countries, exposed to a growing number of ubiquitous chemical substances. It thus increases human exposure pathways: diet, inhalation, soil and dust dermal contact…), notably for semi-volatile organic compounds. Diet is generally sought to contribute the most to total exposure for many chemicals, the relative contribution of each pathway is nevertheless poorly described, and can be different among populations. This is in particularly the case For young children, who can be more exposed via the environment, because of frequent contact with object and dust and hand to mouth behaviors. Children are in addition considered more sensitive to chemical risk due to their maturating systems.

In this context, the objective of this project is to characterize the young children's exposure to a particular class of semi volatile organic compounds. It will encompass the relative contribution of different pathways to the external dose, and to try to match the internal and external doses with a physiologically based pharmacokinetic (PBPK) model for molecules for which it is possible.

The present demand concerns a feasibility study on 2 children, for Perfluorinated Alkylated Substances (PFAS), used in numerous consumer products.

DETAILED DESCRIPTION:
Pilot study for testing feasibility of cross sectional integrative exposure study.

Strategy : Exposure assessment of young children to PFAS with simultaneous measurement of internal (serum) and external doses (diet, indoor environment: contamination data and human exposure factors; quantity ingested and breathed).

Expected outcomes :

Assessment of feasibility to obtain:

* original data on children's body burden
* original contamination data for food, water, air and dust ;
* Matching of these data to identify main sources and pathways of exposure.

ELIGIBILITY:
Inclusion Criteria:

Young children (2-6 months ; 12-18 months)

* In outpatient pediatric or pediatric surgery ;
* From their homes ;
* With home located less than 30km from Rennes ;
* Living at their home (not at childcare facility or child-minder);
* With a scheduled blood sampling apart from this study ;
* For child 2 - 6 months :
* With diet exclusively based on milk (maternal exclusively or commercial exclusively)
* In case of breastfeeding, with mother accepting milk sampling ;
* With a free, enlightened and signed written consent from the parents.

Breastfeeding mother :

* > 18 years ;
* Exclusive breastfeeding ;
* With a free, enlightened and signed written consent.

Exclusion Criteria:

Children :

* Metabolic illness ;
* Renal or hepatic insufficiency ;
* Malabsorption
* With known HIV+, HBV+, HCV+, CMV+ serology
* Simultaneously participating to other biomedical survey

For breastfeeding mother :

* Under legal protection (judicial protection, guardianship) ;
* mixed breastfeeding ;
* with Known HIV+, HBV+, HCV+, CMV+ serology

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Feasibility recruitment | 3 months
  Main objective of this feasibility study is to set the scientific consortium to recruit and study 2 young children's exposures.
  Main judgement criteria : Effective enrolment of 2 young children during their consultation to Rennes hospital, from those having a blood sampling for medical purposes, and house survey.

SECONDARY OUTCOMES:
Protocol validation | 1 year
  Second objective is to validate protocols, procedures and methods to study exposure to PFAS.
  Secondary judgment criteria :
  * Possibility to sample an extra volume of blood, to prepare it and transport it at -18°C to Laberca lab, Nantes;
  * Possibility to organize a home visit with sampling of diet, water, air, dust and delivery of dietary questionnaire;
  * Possibility to quantify PFAS in dietary and environmental samples;
  * Possibility to model the internal dose for some compounds from kinetics data, and to compare doses estimated from blood measurements to those from environmental and diet measurements

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Glorennec, PhD, Study Chair — Inserm UMR 1085 - Institut de Recherche sur la Santé, l'Environnement et le Travail; Florence Rouget, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes Hospital University, Rennes, Brittany Region, France